CLINICAL TRIAL: NCT05130541
Title: Proning Early in Awake COVID-19 Hypoxic Respiratory Failure (PREACHR) Study
Acronym: PREACHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Hospital Queens (Other)
Responsible Party: Principal Investigator, Michael Chary, Instructor, New York Hospital Queens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12910420
Record Dates: First submitted 2021-05-04; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Covid19; Respiratory Failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Non-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Usual Care
  Interventions: Other: Supportive Care
- Proning (Experimental): Proning, rotating 90 degrees on long axis every 30 minutes - 2 hours
  Interventions: Behavioral: Proning; Other: Supportive Care

INTERVENTIONS:
Behavioral: Proning — Rotating on long axis 90 degrees every 30 minutes
  Arms: Proning
Other: Supportive Care — Usual Care

SUMMARY:
The aim of this proposal is to study whether proning, a technique that has previously been shown to improve lung function in patients with acute respiratory distress syndrome (ARDS), can prevent those with mild to moderate symptoms of COVID-19 from progressing to severe disease when initiated early, thereby averting intubation, reducing hospitalization, and, ultimately, decreasing mortality.

DETAILED DESCRIPTION:
COVID-19 is a global pandemic caused by the novel coronavirus SARS-COV-2. At this time, SARS-CoV-2 is believed to infect alveolar cells, directly impairing lung function and eliciting a profound inflammatory response that further damages the lungs. Between 1 in 20 and 1 in 10 patients infected with this virus die.

A crucial decision point in the treatment of patients with COVID-19 in the Emergency Department is the decision to admit to the hospital for further treatment, or discharge the moderately symptomatic (hypoxic and feel ill) but not critically ill patients. However, patients who present with initially mild to moderate symptoms may progress to severe disease. There is, therefore, an unmet need to identify interventions that prevent progression to critical illness in moderately symptomatic patients.

Anecdotal reports from Emergency Physicians suggest that alternating prone and supine positioning (i.e. instructing the patient to periodically turn over) improves hypoxia and delays intubation. Dubbed proning, this technique improves hypoxia in 6-7 out of 10 intubated patients with severe acute respiratory distress syndrome (ARDS). Alternating supine and prone positioning improves the recruitment of alveoli, improves ventilation-perfusion matching, increases end-expiratory lung volumes, and improves pulmonary lymphatic drainage.

This proposal is innovative because it studies the extension of an intervention previously restricted to patients in the intensive care units with severe acute respiratory distress syndrome (ARDS). Current literature on proning in awake patients with ARDS is limited to retrospective studies with no randomized controlled trials. Further, no clinical trials to date have explored the benefits of early awake proning in COVID-19.

The development of a treatment that prevents disease progression and hospitalization in patients moderately ill with COVID-19 would decrease morbidity and mortality from COVID-19 as well as decrease the utilization of scarce healthcare resources. In addition, this trial would be the first randomized controlled-trial, contributing significantly to the nascent evidence base on treatment for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Presenting to the ED with symptoms suggestive of COVID-19
* Assessed by ED attending physician to not require emergent intubation
* Normal mental status and ability to communicate symptoms/distress
* Able to follow instructions independently

Exclusion Criteria:

* Severe respiratory distress requiring immediate intervention
* Unable to follow verbal instructions
* Unable to communicate their needs, symptoms, or distress
* Inability to tolerate prone positioning due to mental status or habitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Within 30 days of discharge from hospital
  All-cause mortality
Need for intubation | At any time during first hospitalization for hypoxia from COVID-19 up to 2 months
  Need for intubation

SECONDARY OUTCOMES:
Number of repeat visits for same complaint | 30 days
  Number of repeat visits in 30 days for same complaint

CONTACTS AND LOCATIONS:
Overall Officials: Richard Shin, MD, Principal Investigator — NYP Queens
Locations (1):
- New York Presbyterian Queens, Flushing, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Will consider compelling cases if appropriately deidentified and, of course, if reviewers or journal editors request
Supporting Information: Study Protocol, SAP, ICF, CSR